CLINICAL TRIAL: NCT01770730
Title: A Randomized Controlled Trial to Evaluate the Impact of Using a Point-of-care Urine LAM Strip Test for TB Diagnosis Amongst Hospitalized HIV-infected Patients in Resource-poor Settings
Brief Title: A Trial of the Urine LAM Strip Test for TB Diagnosis Amongst Hospitalized HIV-infected Patients
Acronym: LAMRCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cape Town (Other)
Collaborators: University of Zimbabwe (Other); University of Zambia (Other); NIMR - Mbeya Medical Research Programme (Unknown)
Responsible Party: Principal Investigator, Jonathan Peter, Honorary consultant, Department of Medicine, University of Cape Town
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: LAMRCT
Record Dates: First submitted 2013-01-11; First posted 2013-01-18 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-06

CONDITIONS: Tuberculosis
Keywords: urine LAM strip test; diagnostics; tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LAM plus standard care (Experimental): Patients allocated to this study arm will receive urine LAM strip testing in addition to the standard TB diagnostic tools WHO approved and available at each site
  Interventions: Device: Urine LAM strip test
- Standard care (No Intervention): Patients allocated to this study arm will receive standard TB diagnostics currently WHO approved and available at the study site

INTERVENTIONS:
Device: Urine LAM strip test — This is a point-of-care lateral flow strip test to detect the presence of lipoarabinomannan (LAM) in patient urine samples. Only patients with a grade 2-5 visual band intensity will be considered positive and commenced on treatment
  Other Names: Determine TB urine LAM Antigen strip test
  Arms: LAM plus standard care

SUMMARY:
The novel urine LAM point-of-care strip test offers potential clinical utility to improve TB diagnosis in HIV co-infected patients. Urine LAM strip test performance improves with increasing illness severity and more advanced immunosuppression, thus offering the greatest potential utility in hospitalised HIV-infected patients with advanced immunosuppression (CD4 cell count less than 200). However, in the context of high rates of empiric treatment and the availability of other novel TB diagnostics, the clinical impact of the urine LAM strip test is unknown. This study will investigate the impact of the urine LAM strip test. The study hypothesis is that the urine LAM strip test, when combined with standard TB diagnostics (smear microscopy and culture) will significantly improve TB treatment-related outcomes (TB-related mortality, morbidity and length of hospital stay) in HIV-infected hospitalized patients when compared to standard TB diagnostics alone.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected (1x rapid HIV test positive)
* Considered TB suspect by attending doctor (must comprise at least 1 of the following: current fever or cough, drenching night sweats, self-reported LOW)
* Illness severity sufficient to warrant hospitalization
* ≥18 years old
* Provision of informed consent

Exclusion Criteria:

* HIV-uninfected
* Patients receiving any anti-TB medication in the 60 days prior to testing
* Unable to provide 30mls urine
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2618 (Actual)
Dates: Start 2013-01; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
All-cause mortality | 8 weeks
  All-cause mortality at 8-weeks after study enrollment

SECONDARY OUTCOMES:
Change in TB-related morbidity score | Baseline and 8 weeks
  Comparative change in TB score between baseline and 8 weeks after enrollment
Change in Karnofsky performance index | Baseline and 8 week
  Comparative changes in the Karnofsky performance index between baseline and 8 weeks following enrollment
Hospital length of stay | Date of hospital discharge (max 8 weeks) minus date of admission
  This is the number of days of hospital admission for enrolled patients up to a maximum of 8 weeks post enrollment.
Diagnostic accuracy of urine LAM strip test | 8 weeks
  Diagnostic accuracy (sensitivity, specificity, predictive values and likelihood ratios) of the urine LAM strip test using TB culture as the diagnostic reference standard

CONTACTS AND LOCATIONS:
Overall Officials: Keertan Dheda, MD, Study Director — UCT Lung Infection and Immunity Unit
Locations (4):
- University of Cape Town, Cape Town, Western Cape, South Africa
- Mbeya Medical Research Programme, Mbeya, Tanzania
- University Teaching Hospital, Lusaka, Zambia
- University of Zimbabwe, Harare, Zimbabwe

REFERENCES:
- [Background] Peter JG, Theron G, van Zyl-Smit R, Haripersad A, Mottay L, Kraus S, Binder A, Meldau R, Hardy A, Dheda K. Diagnostic accuracy of a urine lipoarabinomannan strip-test for TB detection in HIV-infected hospitalised patients. Eur Respir J. 2012 Nov;40(5):1211-20. doi: 10.1183/09031936.00201711. Epub 2012 Feb 23. PMID 22362849
- [Background] Lawn SD, Kerkhoff AD, Vogt M, Wood R. Diagnostic accuracy of a low-cost, urine antigen, point-of-care screening assay for HIV-associated pulmonary tuberculosis before antiretroviral therapy: a descriptive study. Lancet Infect Dis. 2012 Mar;12(3):201-9. doi: 10.1016/S1473-3099(11)70251-1. Epub 2011 Oct 17. PMID 22015305
- [Background] Peter JG, Theron G, Dheda K. Urine antigen test for diagnosis of HIV-associated tuberculosis. Lancet Infect Dis. 2012 Nov;12(11):825; author reply 826-7. doi: 10.1016/S1473-3099(12)70220-7. No abstract available. PMID 23099073
- [Derived] Peter JG, Zijenah LS, Chanda D, Clowes P, Lesosky M, Gina P, Mehta N, Calligaro G, Lombard CJ, Kadzirange G, Bandason T, Chansa A, Liusha N, Mangu C, Mtafya B, Msila H, Rachow A, Hoelscher M, Mwaba P, Theron G, Dheda K. Effect on mortality of point-of-care, urine-based lipoarabinomannan testing to guide tuberculosis treatment initiation in HIV-positive hospital inpatients: a pragmatic, parallel-group, multicountry, open-label, randomised controlled trial. Lancet. 2016 Mar 19;387(10024):1187-97. doi: 10.1016/S0140-6736(15)01092-2. Epub 2016 Mar 10. PMID 26970721